CLINICAL TRIAL: NCT00195273
Title: A Randomized Open-Label Study Comparing the Efficacy and Safety of Sirolimus Combined With Daclizumab, Mycophenolate and Corticosteroids vs Cyclosporine, Mycophenolate and Corticosteroids in Renal Allograft Recipients Receiving Kidneys From Older Donors
Brief Title: Study Evaluating Sirolimus in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H-101466
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Graft vs Host Disease; Kidney Transplantation
Keywords: Kidney; Transplant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus; Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sirolimus + Daclizumab + Mycophenolate + Corticosteroids
  Interventions: Drug: sirolimus; Drug: mycophenolate mofetil; Drug: corticosteroids; Drug: daclizumab
- 2 (Active Comparator): Cyclosporine + Mycophenolate + Corticosteroids
  Interventions: Drug: cyclosporine; Drug: mycophenolate mofetil; Drug: corticosteroids

INTERVENTIONS:
Drug: sirolimus — 15 mg loading dose, followed by 5 mg/day to achieve target trough levels of 10-15 ng/mL at months 1-6, then 8-12 ng/mL at months 7-12
  Arms: 1
Drug: cyclosporine — Initial dose of 10 mg/kg/day, then twice daily to achieve target trough levels of 300-400 ng/mL at weeks 0-4; 200-300 ng/mL at months 1-2; 150-250 ng/mL at months 2-3; 100-200 ng/mL at months 3-6; 75-150 ng/mL months 6-12
  Arms: 2
Drug: mycophenolate mofetil — 1 g twice daily; may be reduced to 750 mg BID for adverse events, or to 500 mg BID for persisting adverse events
Drug: corticosteroids — As per center practice. By day 8 prednisolone tapered to 20 mg/day; by day 30 to 15 mg/day; by day 60 to 10 mg/day; after 4 to 6 months to 5-7.5 mg/day
Drug: daclizumab — IV: 1 mg/kg to a maximum of 100 mg/dose. 5 doses at 2, 4, 6, and 8 weeks after transplantation
  Arms: 1

SUMMARY:
The purpose of this study is to compare the kidney function in patients who have received a transplanted kidney and were treated with the combination of sirolimus, daclizumab, mycophenolate and corticosteroids versus transplanted patients treated with cyclosporine, mycophenolate and corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation
* Donor must be at least 60 years old.

Exclusion Criteria:

* Current systemic infection
* Unstable angina or treatment for serious arrhythmia.
* Cancer within the previous 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Norway, Sweden, MedInfoNord@wyeth.com
Locations (3):
- Oslo, Norway
- Sweden (2):
  - Gothenburg
  - Uppsala

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Sweden from November 2004 to September 2007.
Pre-assignment Details: Prior to enrollment in study, patients were screened for eligibility. If eligibility criteria were met, patients were enrolled and randomized.
Groups:
- Sirolimus: Sirolimus: initiated within 24 hours before or after transplantation; Loading dose of 15mg followed by 5mg/day (morning) until doses are adjusted to achieve steady state whole-blood trough levels of 10-15ng/ml during months 1-6, followed by 8-12ng/ml during months 7-12 Daclizumab: administered intravenously over 15 minutes at a dose of 1mg/kg to a maximum of 100mg per dose. First dose administered within24 hours before transplantation, with subsequent doses at weeks 2, 4, 6 and 8 weeks after transplantation, for a total of five doses.
  Mycophenolate mofetil: 1000mg twice daily. Dose can be reduced to 750mg twice daily in the case of adverse events and reduced further to 500mg if adverse events persist.
  Corticosteroids: given according to transplant center standard of care pre- and postoperatively. By day 8 prednisolone should be tapered to 20mg/day, by day 30 to 15mg/day, by day 60 to 10mg/day, and after 4-6 months to 5-7.5mg/day.
- Cyclosporine (CsA): Cyclosporine: first dose of 10mg/kg/day administered orally or via a NG-tube, no later than 24 hours after transplant. (First dose may be initiated prior to transplantation.) Subsequent doses given in equally divided doses (where possible) of twice daily at approximately 12-hour intervals. The subsequent doses should be adjusted to achieve target therapeutic ranges in whole blood.
  Mycophenolate mofetil: 1000mg twice daily. Dose can be reduced to 750mg twice daily in the case of adverse events and reduced further to 500mg if adverse events persist.
  Corticosteroids: given according to transplant center standard of care pre- and postoperatively. By day 8 prednisolone should be tapered to 20mg/day, by day 30 to 15mg/day, by day 60 to 10mg/day, and after 4-6 months to 5-7.5mg/day.
Period: Overall Study
Arm/Group | Sirolimus | Cyclosporine (CsA)
Started | 31 | 30
Completed | 10 | 16
Not Completed | 21 | 14
Not completed — Adverse Event | 9 | 9
Not completed — Protocol deviation | 0 | 1
Not completed — Lack of Efficacy | 3 | 1
Not completed — Procedural complications | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Cyclosporine (CsA) | Total
Number analyzed (Participants) | 31 | 30 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 61.00 (10.00) | 59.60 (10.10) | 60.31 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Creatinine Clearance Rate
Description: Creatinine clearance is a measure of kidney function. Creatinine clearance rate is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Creatinine clearance can be measured directly or estimated using established formulas. For this study, the creatinine clearance rate was calculated using the Nankivell formula. Normal values for healthy, young males are in the range of 100-135 ml/min and for females 90-125 ml/min. A low creatinine clearance indicates poor kidney function.
Time Frame: 12 months
Population: All patients who completed 12 months of study drug.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Sirolimus | Cyclosporine (CsA)
Number analyzed (Participants) | 20 | 20
ml/min | 56.800 (21.522) | 53.449 (15.497)
Statistical Analysis 1: Comparison: Sirolimus vs Cyclosporine (CsA); Test type: Superiority or Other; p = 0.6081, ANOVA — Calculated for 12 month analysis; Analysis of variance with treatment group and center as factors

2. Secondary Outcome: Number of Patients With Acute Rejection
Description: The diagnosis of acute rejection was made via kidney biopsy (Banff criteria). The Banff criteria are standardized diagnostic categories based on histological assessments (e.g., cell types and distributions). Biopsy was performed before initiation of anti-rejection therapy, or at least within 24 hours of the start of therapy.
Time Frame: 3 and 12 months
Population: All patients who received at least one dose of study drug.
Measure: Number; unit: patients
Arm/Group | Sirolimus | Cyclosporine (CsA)
Number analyzed (Participants) | 31 | 30
patients
  3 months | 3 | 9
  12 months | 5 | 10

3. Secondary Outcome: Patient and Graft Survival
Description: Graft survival is measured by graft loss which is defined as removal of the transplant.
Time Frame: 12 months
Population: All patients who received at least one dose of study drug.
Measure: Number; unit: patients
Arm/Group | Sirolimus | Cyclosporine (CsA)
Number analyzed (Participants) | 31 | 30
patients
  Patient survival | 31 | 29
  Graft loss | 0 | 3

4. Secondary Outcome: Mean Creatinine Clearance Rate - 3 Months
Description: as for outcome 1
Time Frame: 3 months
Population: All patients who completed 3 months of study drug.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Sirolimus | Cyclosporine (CsA)
Number analyzed (Participants) | 27 | 27
ml/min | 55.200 (22.403) | 51.878 (15.974)
Statistical Analysis 1: Comparison: Sirolimus vs Cyclosporine (CsA); Test type: Superiority or Other; p = 0.4662, ANOVA; Calculated for 3 month analysis

ADVERSE EVENTS:
Arm/Group | Sirolimus | Cyclosporine (CsA)
Serious Adverse Events (participants affected / at risk) | 26 | 24
Other Adverse Events (participants affected / at risk) | 31 | 30
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sirolimus | Cyclosporine (CsA)
Anemia (Blood and lymphatic system disorders) | 2/31 | 2/30
Lymphocele (Blood and lymphatic system disorders) | 4/31 | 6/30
Atrial fibrillation (Cardiac disorders) | 1/31 | 1/30
Myocardial infarction (Cardiac disorders) | 1/31 | 0/30
Abdominal pain (Gastrointestinal disorders) | 0/31 | 1/30
Anal hemorrhage (Gastrointestinal disorders) | 1/31 | 0/30
Constipation (Gastrointestinal disorders) | 0/31 | 1/30
Diarrhea (Gastrointestinal disorders) | 0/31 | 1/30
Gastritis (Gastrointestinal disorders) | 0/31 | 1/30
Hemorrhoids (Gastrointestinal disorders) | 1/31 | 0/30
Ileus (Gastrointestinal disorders) | 0/31 | 1/30
Melaena (Gastrointestinal disorders) | 1/31 | 0/30
General malaise (General disorders) | 1/31 | 0/30
Hernia (General disorders) | 2/31 | 0/30
Oedema (General disorders) | 1/31 | 0/30
Pyrexia (General disorders) | 0/31 | 1/30
Cholecystitis acute (Hepatobiliary disorders) | 0/31 | 1/30
Kidney transplant rejection (Immune system disorders) | 4/31 | 8/30
Transplant rejection (Immune system disorders) | 0/31 | 2/30
Brain abscess (Infections and infestations) | 0/31 | 1/30
Cystitis (Infections and infestations) | 0/31 | 2/30
Cytomegalovirus infection (Infections and infestations) | 3/31 | 5/30
Diverticulitis (Infections and infestations) | 0/31 | 1/30
Ear infection (Infections and infestations) | 0/31 | 1/30
Escherichia sepsis (Infections and infestations) | 1/31 | 0/30
Gastroenteritis (Infections and infestations) | 1/31 | 0/30
Pneumonia (Infections and infestations) | 3/31 | 4/30
Pneumonia cytomegaloviral (Infections and infestations) | 1/31 | 0/30
Sepsis (Infections and infestations) | 1/31 | 1/30
Upper respiratory tract infection (Infections and infestations) | 1/31 | 0/30
Urinary tract infection (Infections and infestations) | 3/31 | 0/30
Urosepsis (Infections and infestations) | 0/31 | 1/30
Varicella (Infections and infestations) | 0/31 | 1/30
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1/31 | 0/30
Graft thrombosis (Injury, poisoning and procedural complications) | 0/31 | 1/30
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1/31 | 0/30
Renal graft loss (Injury, poisoning and procedural complications) | 0/31 | 1/30
Subdural haematoma (Injury, poisoning and procedural complications) | 0/31 | 1/30
Upper limb fracture (Injury, poisoning and procedural complications) | 0/31 | 1/30
Wound complication (Injury, poisoning and procedural complications) | 3/31 | 0/30
Wound dehiscence (Injury, poisoning and procedural complications) | 2/31 | 0/30
Wound hemorrhage (Injury, poisoning and procedural complications) | 0/31 | 1/30
Blood creatinine increased (Investigations) | 1/31 | 3/30
Fluid retention (Metabolism and nutrition disorders) | 1/31 | 0/30
Hyponatraemia (Metabolism and nutrition disorders) | 0/31 | 1/30
Back pain (Musculoskeletal and connective tissue disorders) | 0/31 | 1/30
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/31 | 1/30
Myalgia (Musculoskeletal and connective tissue disorders) | 1/31 | 0/30
Epilepsy (Nervous system disorders) | 0/31 | 1/30
Transient ischaemic attack (Nervous system disorders) | 0/31 | 1/30
Bladder disorder (Renal and urinary disorders) | 0/31 | 1/30
Glomerulonephritis (Renal and urinary disorders) | 0/31 | 1/30
Hydronephrosis (Renal and urinary disorders) | 1/31 | 1/30
Renal artery stenosis (Renal and urinary disorders) | 1/31 | 1/30
Renal impairment (Renal and urinary disorders) | 3/31 | 1/30
Ureteric obstruction (Renal and urinary disorders) | 0/31 | 1/30
Ureteric stenosis (Renal and urinary disorders) | 1/31 | 1/30
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Aneurysm (Vascular disorders) | 1/31 | 0/30
Hematoma (Vascular disorders) | 1/31 | 0/30
Hemorrhage (Vascular disorders) | 0/31 | 1/30
Transplant changes (General disorders) | 0/31 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sirolimus | Cyclosporine (CsA)
Anemia (Blood and lymphatic system disorders) | 15/31 | 17/30
Leukopenia (Blood and lymphatic system disorders) | 4/31 | 7/30
Lymphocele (Blood and lymphatic system disorders) | 3/31 | 3/30
Arrhythmia (Cardiac disorders) | 9/31 | 6/30
Atrial fibrillation (Cardiac disorders) | 0/31 | 1/30
Bradycardia (Cardiac disorders) | 6/31 | 3/30
Palpitations (Cardiac disorders) | 1/31 | 1/30
Sinus tachycardia (Cardiac disorders) | 1/31 | 1/30
Tachycardia (Cardiac disorders) | 0/31 | 1/30
Hydrocele (Congenital, familial and genetic disorders) | 0/31 | 1/30
Cerumen impaction (Ear and labyrinth disorders) | 0/31 | 1/30
Deafness (Ear and labyrinth disorders) | 0/31 | 1/30
Ear pain (Ear and labyrinth disorders) | 1/31 | 0/30
Hyperaldosteronism (Endocrine disorders) | 0/31 | 1/30
Eye edema (Eye disorders) | 1/31 | 0/30
Visual acuity reduced (Eye disorders) | 2/31 | 1/30
Abdominal pain (Gastrointestinal disorders) | 0/31 | 3/30
Constipation (Gastrointestinal disorders) | 4/31 | 7/30
Diarrhea (Gastrointestinal disorders) | 7/31 | 2/30
Dry mouth (Gastrointestinal disorders) | 2/31 | 0/30
Duodenal ulcer (Gastrointestinal disorders) | 1/31 | 0/30
Dyspepsia (Gastrointestinal disorders) | 1/31 | 1/30
Flatulence (Gastrointestinal disorders) | 0/31 | 1/30
Gastritis (Gastrointestinal disorders) | 1/31 | 3/30
Gastrointestinal disorder general (Gastrointestinal disorders) | 1/31 | 1/30
Gingival hyperplasia (Gastrointestinal disorders) | 0/31 | 2/30
Gingivitis (Gastrointestinal disorders) | 0/31 | 1/30
Hemorrhodial hemorrhage (Gastrointestinal disorders) | 1/31 | 0/30
Hemorrhoids (Gastrointestinal disorders) | 3/31 | 2/30
Hypoaesthesia oral (Gastrointestinal disorders) | 0/31 | 1/30
Intra-abdominal hematoma (Gastrointestinal disorders) | 1/31 | 0/30
Lip ulceration (Gastrointestinal disorders) | 1/31 | 0/30
Melaena (Gastrointestinal disorders) | 0/31 | 2/30
Nausea (Gastrointestinal disorders) | 7/31 | 10/30
Esophagitis (Gastrointestinal disorders) | 0/31 | 1/30
Gastric refulx (Gastrointestinal disorders) | 0/31 | 1/30
Stomach discomfort (Gastrointestinal disorders) | 0/31 | 1/30
Stomatitis (Gastrointestinal disorders) | 1/31 | 0/30
Tongue ulceration (Gastrointestinal disorders) | 1/31 | 0/30
Vomiting (Gastrointestinal disorders) | 1/31 | 2/30
Calcinosis (General disorders) | 0/31 | 1/30
Chest pain (General disorders) | 1/31 | 1/30
Chills (General disorders) | 1/31 | 2/30
Discomfort (General disorders) | 1/31 | 0/30
Fatigue (General disorders) | 1/31 | 2/30
Feeling abnormal (General disorders) | 1/31 | 0/30
Feeling cold (General disorders) | 0/31 | 1/30
Fibrosis (General disorders) | 0/31 | 1/30
Hernia (General disorders) | 1/31 | 1/30
Impaired healing (General disorders) | 4/31 | 1/30
Malaise (General disorders) | 1/31 | 0/30
Necrosis (General disorders) | 1/31 | 0/30
Oedema (General disorders) | 8/31 | 4/30
Adema peripheral (General disorders) | 10/31 | 9/30
Pyrexia (General disorders) | 3/31 | 2/30
Vessel puncture site hemorrhage (General disorders) | 0/31 | 1/30
Hypersenstivity (Immune system disorders) | 0/31 | 1/30
Kidney transplant rejection (Immune system disorders) | 3/31 | 8/30
Transplant rejection (Immune system disorders) | 0/31 | 1/30
Anogenital warts (Infections and infestations) | 0/31 | 1/30
Asymptomatic bacteriuria (Infections and infestations) | 0/31 | 1/30
Bronchitis (Infections and infestations) | 4/31 | 1/30
Candidiasis (Infections and infestations) | 0/31 | 1/30
Candiduria (Infections and infestations) | 0/31 | 1/30
Citrobacter infection (Infections and infestations) | 1/31 | 0/30
Clostridial infection (Infections and infestations) | 1/31 | 0/30
Cystitis (Infections and infestations) | 4/31 | 4/30
Cytomegalovirus infection (Infections and infestations) | 3/31 | 6/30
Ear infection (Infections and infestations) | 1/31 | 0/30
Escherichia urinary tract infection (Infections and infestations) | 0/31 | 1/30
Folliculitis (Infections and infestations) | 1/31 | 0/30
Fungal infection (Infections and infestations) | 0/31 | 1/30
Genital infection fungal (Infections and infestations) | 0/31 | 1/30
Herpes simplex (Infections and infestations) | 2/31 | 2/30
Herpes virus infection (Infections and infestations) | 1/31 | 2/30
Herpes zoster (Infections and infestations) | 0/31 | 2/30
Human polyomavirus (Infections and infestations) | 1/31 | 0/30
Infection (Infections and infestations) | 2/31 | 1/30
Viral laryngitis (Infections and infestations) | 0/31 | 1/30
Nasopharyngitis (Infections and infestations) | 4/31 | 4/30
Oral candidiasis (Infections and infestations) | 4/31 | 2/30
Oral fungal infection (Infections and infestations) | 1/31 | 1/30
Oral herpes (Infections and infestations) | 1/31 | 0/30
Orchitis (Infections and infestations) | 1/31 | 0/30
Pharyngitis (Infections and infestations) | 0/31 | 1/30
Pneumonia (Infections and infestations) | 3/31 | 0/30
Postoperative wound infection (Infections and infestations) | 1/31 | 0/30
Sepsis (Infections and infestations) | 0/31 | 1/30
Sinusitis (Infections and infestations) | 1/31 | 1/30
Transplant failure (Infections and infestations) | 0/31 | 1/30
Upper respiratory tract infection (Infections and infestations) | 0/31 | 1/30
Urinary tract infection (Infections and infestations) | 8/31 | 4/30
Wound infection (Infections and infestations) | 0/31 | 1/30
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2/31 | 2/30
Drug toxicity (Injury, poisoning and procedural complications) | 2/31 | 0/30
Excoriation (Injury, poisoning and procedural complications) | 1/31 | 1/30
Fall (Injury, poisoning and procedural complications) | 1/31 | 1/30
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1/31 | 0/30
Postoperative wound complication (Injury, poisoning and procedural complications) | 3/31 | 1/30
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1/31 | 0/30
Tracheal obstruction (Injury, poisoning and procedural complications) | 0/31 | 1/30
Wound (Injury, poisoning and procedural complications) | 1/31 | 1/30
Wound complications (Injury, poisoning and procedural complications) | 0/31 | 1/30
Alanine aminotransferase increased (Investigations) | 1/31 | 0/30
Antibody test positive (Investigations) | 0/31 | 1/30
Blood creatinine increased (Investigations) | 3/31 | 3/30
Blood glucose increased (Investigations) | 3/31 | 2/30
Blood magnesium decreased (Investigations) | 0/31 | 1/30
Blood parathyroid hormone (Investigations) | 0/31 | 1/30
Blood potassium increased (Investigations) | 1/31 | 0/30
Blood urea increased (Investigations) | 0/31 | 1/30
Blood uric acid increased (Investigations) | 0/31 | 1/30
C-reactive protein increased (Investigations) | 1/31 | 1/30
Cardiac murmur (Investigations) | 2/31 | 1/30
Cytomegalovirus test postive (Investigations) | 0/31 | 2/30
Hepatic enzyme increased (Investigations) | 1/31 | 0/30
Transaminases increased (Investigations) | 1/31 | 1/30
Weight increased (Investigations) | 2/31 | 0/30
Diabetes mellitus (Metabolism and nutrition disorders) | 6/31 | 1/30
Food intolerance (Metabolism and nutrition disorders) | 0/31 | 1/30
Hypercalcaemia (Metabolism and nutrition disorders) | 1/31 | 1/30
Hypercholesterolemia (Metabolism and nutrition disorders) | 0/31 | 2/30
Hyperglycemia (Metabolism and nutrition disorders) | 0/31 | 1/30
Hyperkalaemia (Metabolism and nutrition disorders) | 3/31 | 3/30
Hyperlipidaemia (Metabolism and nutrition disorders) | 4/31 | 2/30
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1/31 | 1/30
Hypocalcaemia (Metabolism and nutrition disorders) | 2/31 | 2/30
Hypokalaemia (Metabolism and nutrition disorders) | 1/31 | 2/30
Hyponatraemia (Metabolism and nutrition disorders) | 0/31 | 2/30
Hypophosphataemia (Metabolism and nutrition disorders) | 1/31 | 0/30
Malnutrition (Metabolism and nutrition disorders) | 1/31 | 0/30
Metabolic acidosis (Metabolism and nutrition disorders) | 2/31 | 0/30
Podagra (Metabolism and nutrition disorders) | 0/31 | 1/30
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/31 | 1/30
Back pain (Musculoskeletal and connective tissue disorders) | 1/31 | 3/30
Fistula (Musculoskeletal and connective tissue disorders) | 1/31 | 0/30
Groin pain (Musculoskeletal and connective tissue disorders) | 0/31 | 1/30
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1/31 | 0/30
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/31 | 1/30
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/31 | 1/30
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/31 | 0/30
Myalgia (Musculoskeletal and connective tissue disorders) | 1/31 | 1/30
Osteitis (Musculoskeletal and connective tissue disorders) | 1/31 | 0/30
Osteopenia (Musculoskeletal and connective tissue disorders) | 3/31 | 1/30
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2/31 | 1/30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/31 | 1/30
Tendon pain (Musculoskeletal and connective tissue disorders) | 0/31 | 1/30
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/31 | 0/30
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/31 | 2/30
Dizziness (Nervous system disorders) | 0/31 | 1/30
Dizziness postural (Nervous system disorders) | 2/31 | 0/30
Epilepsy (Nervous system disorders) | 0/31 | 1/30
Headache (Nervous system disorders) | 2/31 | 1/30
Metabolic encephalopathy (Nervous system disorders) | 1/31 | 0/30
Paraesthesia (Nervous system disorders) | 0/31 | 1/30
Peroneal nerve palsy (Nervous system disorders) | 0/31 | 2/30
Sciatica (Nervous system disorders) | 0/31 | 1/30
Sensory loss (Nervous system disorders) | 0/31 | 1/30
Syncope (Nervous system disorders) | 0/31 | 1/30
Tremor (Nervous system disorders) | 0/31 | 2/30
Confusional state (Psychiatric disorders) | 1/31 | 2/30
Depressed mood (Psychiatric disorders) | 0/31 | 1/30
Insomina (Psychiatric disorders) | 2/31 | 0/30
Nightmare (Psychiatric disorders) | 0/31 | 1/30
Anuria (Renal and urinary disorders) | 0/31 | 1/30
Bladder stenosis (Renal and urinary disorders) | 0/31 | 1/30
Hematuria (Renal and urinary disorders) | 3/31 | 2/30
Hydronephrosis (Renal and urinary disorders) | 0/31 | 1/30
Nocturia (Renal and urinary disorders) | 1/31 | 0/30
Oliguria (Renal and urinary disorders) | 1/31 | 1/30
Proteinuria (Renal and urinary disorders) | 2/31 | 0/30
Renal impairment (Renal and urinary disorders) | 0/31 | 1/30
Renal tubular necrosis (Renal and urinary disorders) | 1/31 | 0/30
Erectile dysfunction (Reproductive system and breast disorders) | 0/31 | 1/30
Testicular pain (Reproductive system and breast disorders) | 0/31 | 1/30
Vaginal discharge (Reproductive system and breast disorders) | 1/31 | 0/30
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/31 | 1/30
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Cough (Respiratory, thoracic and mediastinal disorders) | 4/31 | 5/30
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/31 | 1/30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3/31 | 2/30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4/31 | 0/30
Nasal conjestion (Respiratory, thoracic and mediastinal disorders) | 1/31 | 1/30
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0/31 | 1/30
Obstructive airway disorder (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0/31 | 1/30
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0/31 | 1/30
Snoring (Respiratory, thoracic and mediastinal disorders) | 1/31 | 0/30
Acne (Skin and subcutaneous tissue disorders) | 1/31 | 1/30
Angioedema (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0/31 | 1/30
Dermatitis (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Eczema (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Hidradenitis (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Hirsutism (Skin and subcutaneous tissue disorders) | 1/31 | 2/30
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/31 | 1/30
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0/31 | 1/30
Night sweats (Skin and subcutaneous tissue disorders) | 1/31 | 1/30
Petechiae (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Pruritus (Skin and subcutaneous tissue disorders) | 0/31 | 2/30
Rash (Skin and subcutaneous tissue disorders) | 1/31 | 2/30
Rash erythematous (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Skin irritation (Skin and subcutaneous tissue disorders) | 0/31 | 1/30
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Swelling face (Skin and subcutaneous tissue disorders) | 0/31 | 1/30
Urticaria (Skin and subcutaneous tissue disorders) | 1/31 | 0/30
Renal surgery (Surgical and medical procedures) | 1/31 | 0/30
Urethral operation (Surgical and medical procedures) | 0/31 | 1/30
Angiodysplasia (Vascular disorders) | 1/31 | 0/30
Deep vein thrombosis (Vascular disorders) | 1/31 | 0/30
Haematoma (Vascular disorders) | 4/31 | 1/30
Hemorrhage (Vascular disorders) | 1/31 | 1/30
Hypertension (Vascular disorders) | 4/31 | 2/30
Injection site reaction (General disorders) | 1/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.